CLINICAL TRIAL: NCT06542081
Title: The Effect of Psychological Resilience Levels of Parents With Hearing Impaired Children on Disaster Preparedness
Brief Title: Psychological Resilience and Disaster Preparedness
Acronym: disaster
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Abdullah Adiyaman, Graduate Student, Yuzuncu Yil University
Other Study IDs: YuzuncıYıl 3
Record Dates: First submitted 2024-08-01; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Psychological Resilience and Disaster Preparedness
Keywords: Disaster Preparedness; Psychological Resilience; Hearing Impaired Children; Parents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One grup: parents of hearing impaired children
  Interventions: Behavioral: Descriptive information form, psychological resilience scale and disaster preparedness scale were completed by the parents of hearing impaired children.

INTERVENTIONS:
Behavioral: Descriptive information form, psychological resilience scale and disaster preparedness scale were completed by the parents of hearing impaired children. — Descriptive information form, psychological resilience scale and disaster preparedness scale were completed by the parents of hearing impaired children.

SUMMARY:
Given our geographical location, there is always the possibility of encountering a disaster at any moment. It is a well-known fact that families with children who have special needs face a series of challenges throughout their lives, and these challenges are known to increase during disaster situations. Therefore, it is emphasized that families with children who have special needs should be supported in every aspect. This study aims to examine the relationship between the psychological resilience levels of parents with hearing-impaired children and their disaster preparedness. With this research, the question "How can the relationship between the psychological resilience levels of parents with hearing-impaired children and their disaster preparedness be assessed, and can this relationship provide insights into how more effective support can be provided to families?" seeks an answer.

DETAILED DESCRIPTION:
Hearing plays crucial roles in communication, responding to environmental stimuli, ensuring safety, and increasing environmental awareness. Hearing impairment refers to the partial or complete loss of a person's hearing ability. Individuals with hearing impairment experience hearing or understanding difficulties differently from those with normal hearing abilities. The degree and effects of hearing impairment vary from person to person and can be congenital or acquired later in life. Congenital hearing impairment is often due to genetic or prenatal factors, while acquired hearing loss can result from various factors such as diseases, accidents, and infections.

Throughout their lives, individuals encounter numerous adverse, traumatic, anxious, and stressful events. The ability to recover and quickly return to normal life after such experiences is explained by the concept of psychological resilience in positive psychology. Psychological resilience, as defined by the American Psychiatric Association, is the ability to adapt, recover, and effectively cope with significant issues such as traumas, serious health problems, and financial difficulties.

Disaster preparedness plays a significant role in reducing losses and destruction in all disaster situations. Preparedness is closely related to the concepts of risk, threat, and vulnerability. Effective disaster preparedness plans are particularly critical for children with disabilities, who are especially vulnerable during disasters. Enhanced preparedness can mitigate the care disruptions that arise during disasters, and better planning can reduce the negative responses to disaster-related stress factors.

Parents of children with disabilities face high caregiving burdens and psychological challenges even without disasters. Studies show that these parents often experience feelings of frustration, helplessness, anger, and depression, highlighting the need for psychological support and relief from caregiving burdens. Effective family preparation plans and targeted education can benefit parents of developmentally disabled children, providing opportunities and methods for public health and safety planning, education, and access.

Resilience interventions supporting parents of children with cancer and other special needs have shown positive effects, including enhanced social connections and support among parents.Studies indicate that parents' levels of self-compassion, psychological resilience, and social support significantly impact their overall well-being.

Literature reviews reveal that studies often focus on the psychological resilience levels of parents with mentally disabled children, with findings emphasizing the need for support. However, there is a lack of research specifically examining the psychological resilience levels of parents with hearing-impaired children. This study aims to address this gap by evaluating the psychological resilience and disaster preparedness levels of parents with hearing-impaired children, thereby contributing valuable insights into how to assess resilience and preparedness for different disability groups.

ELIGIBILITY:
Inclusion Criteria:

* With a hearing-impaired child,
* 21-48 years old,
* open to communication,
* voluntary participation in the study,
* parents without any disability to participate in the study

Exclusion Criteria:

* No hearing impaired children,
* closed to communication,
* who do not accept voluntary participation in the study,
* parents with any disability

Ages: 21 Years to 48 Years | Sex: All
Age Groups: Adult
Study Population: parents with hearing impaired children
Sampling Method: Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-14 (Actual)

PRIMARY OUTCOMES:
psychological resilience scale | 6 monts
  The scale consists of a total of 21 items. It is rated on a five-point Likert scale ranging from "Completely describes me (5)" to "Does not describe me at all (1)." Higher scores indicate higher psychological resilience. The scale comprises four sub-dimensions: Relational Resources, Individual Resources, Cultural and Contextual Resources, and Familial Resources.
disaster preparedness scale | 6 monts
  The Disaster Preparedness Scale consists of 15 questions and 4 sub-dimensions. The four factors are named as follows: Disaster Physical Protection (DPP), Planning (P), Disaster Aid (DA), and Disaster Warning and Signals (DWS). The DPP factor consists of 7 items with factor loadings ranging from .79 to .40; The P factor consists of 3 items with factor loadings ranging from .84 to .75;. The DA factor consists of 3 items with factor loadings ranging from .78 to .60.
Descriptive information form | 6 monts
  Based on the literature, a 23-question form has been created to determine socio-demographic characteristics such as age, gender, income status, presence of chronic illness, number of children, and the place where the family lives.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Adıyaman, Principal Investigator — abdullah.adiyaman@erzurum.edu.tr
Locations (1):
- Van Yuzuncu Yıl University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No